CLINICAL TRIAL: NCT02384590
Title: Feasibility of Implementing Mental Health Treatment in Routine Adult Sickle Cell Disease Care Using Online Cognitive Behavioral Therapy and a Mobile Technology-Based Intervention
Brief Title: Cognitive Behavioral Therapy and Real-time Self-management Intervention for SCD Via Mobile Applications
Acronym: CaRISMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Charles Jonassaint, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO14120495
Record Dates: First submitted 2015-02-26; First posted 2015-03-10 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Sickle Cell Disease; Depression; Anxiety
MeSH Terms: conditions — Anemia, Sickle Cell; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CCBT + Care Manager Arm (Experimental): Patients will be given a tablet device with unlimited data. The device will be pre-installed with a pain and mood diary app that will prompt them to enter their pain severity (0-10), pain location, and mood (0-10), once a day. They will also be registered on to the Beating the Blues website and asked to use the tablet device to complete eight 1-hour Beating the Blues CBT sessions, over the next 3-months. They will also be introduced to a care manager who will contact them on a weekly basis by telephone and throughout the week by email or text, for one-month and then as needed for two additional months. At the conclusion of 3 months participants will only have care manager support upon request but are free to continue using the Beating the Blues program for as long as they like.
  Interventions: Behavioral: Computerized cognitive behavioral therapy
- Treatment As Usual (No Intervention): Similar to the treatment arm, patients will be given a tablet device with unlimited data that comes pre-loaded with a pain and mood diary app. The app will prompt the usual care patients to complete diary data daily. No other activities are required as part of the study but the patients are free to use the tablet as much as they like for their own leisure. At the end of 3-months, patients who continue to report depressive or anxiety symptoms are invited to cross-over to the treatment arm where they will be registered for the Beating the Blues program and given care manger support.

INTERVENTIONS:
Behavioral: Computerized cognitive behavioral therapy — The "Beating the Blues" computerized cognitive behavioral therapy (CCBT) program is eight 50-minute online sessions that teach the participant how to better manage stress using cognitive behavioral therapy techniques. Cognitive behavioral therapy involves helping people change their thoughts and behaviors so they can limit the negative impact stress will have on their mood and pain experience.
  Other Names: online cognitive behavioral therapy; Internet-delivered cognitive behavioral therapy; Beating the Blues
  Arms: CCBT + Care Manager Arm

SUMMARY:
Patients with sickle cell disease (SCD) experience significant depressive symptoms that currently go unrecognized and under-treated. Further, depression in this patient population has the potential to contribute to high health care utilization and poor disease outcomes; however, there are currently no comparative effectiveness studies of evidenced-based mental health treatments for depression in SCD.

The primary objective of this study is to test the effectiveness of an online computerized cognitive behavioral therapy intervention to address psychological and behavioral needs of patients with sickle cell disease, namely depression and pain symptoms. The investigators will implement an existing computerized cognitive behavioral therapy (CCBT) program called "Beating the Blues" into routine clinical care at the University of Pittsburgh Medical Center (UPMC) Adult Sickle Cell Clinic to determine the effectiveness of this intervention in decreasing depression and pain versus treatment as usual. Patients with significant distress-depression and/or anxiety symptoms-will be randomized to either eight sessions of a CCBT program and weekly follow-up with a care manager or treatment as usual where the treating physician is notified of the patient's symptoms. The investigators will evaluate patient acceptability, implementation and practicality of the online mental health intervention through patient use of the site (frequency and duration of visits), qualitative interviews, and surveys. The investigators hypothesize: 1) the CCBT will be an acceptable mental health treatment for patients and easily integrated into routine clinical care; 2) patients in the treatment arm will show a greater decrease in depression/anxiety symptoms and average daily pain than patients in usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at baseline visit.
2. Documentation of a SCD diagnosis (HgbSS, HgbSC, SBeta +Thal; or SBeta oThal)
3. Receive routine care at the UPMC sickle cell clinic.
4. Scores indicative of clinically significant depression or anxiety on the stress/pain screener that is administered as part of routine SCD care to all patients. i.e. Patient Health Questionnaire (PHQ-9) ≥ 10 and/or Generalized Anxiety Disorder scale (GAD-7) ≥ 8

Exclusion Criteria:

1. Presence of a condition or abnormality (e.g. significant neurocognitive dysfunction) that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Patient acceptability as measured by CCBT sessions completed | 6-months
  Number of CCBT sessions completed while enrolled in study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States